CLINICAL TRIAL: NCT04139369
Title: Study of DNA Methylation in Children and Adolescents With Type 1 Diabetes Mellitus
Brief Title: Methylation of DNA in Children and Adolescents With Type 1 Diabetes Mellitus (METHYLDIAB)
Acronym: METHYLDIAB
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Assimina Galli-Tsinopoulou, PROFESSOR, Aristotle University Of Thessaloniki
Other Study IDs: PEDIATRIC DIABETOLOGY
Record Dates: First submitted 2016-01-09; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: INS gene; methylation; next generation sequencing
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Insulin-Dependent, 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA from white blood cells from peripheral blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 Diabetes Mellitus (T1DM): Type 1 Diabetes Mellitus (T1DM) Children and adolescents with Type 1 Diabetes Mellitus
- Controls (C): Controls (C) Healthy individuals matched for gender and age without any autoimmune disease of their own or their first degree relatives

SUMMARY:
Type 1 Diabetes Mellitus (T1DM) is a well-studied autoimmune disease resulting in insulin deficiency due to selective β-cell destruction. Epigenetics is a novel field of biology studying the inherited changes in deoxyribonucleic acid (DNA) expression which cannot be attributed to base sequence alteration. A relatively limited number of studies are published until now concerning T1DM in children and adolescents addressing epigenetics changes in DNA expression. The purpose of the present study is to analyze the methylation status of DNA within the promoter region of specific susceptibility genes such as Protein tyrosine phosphatase, non-receptor type 22 (PTPN-22), Insulin (INS) and Human leukocyte antigen G (HLA-G) genes.

DETAILED DESCRIPTION:
Type 1 Diabetes Mellitus (T1DM) is a well-studied autoimmune disease resulting in insulin deficiency due to selective β-cell loss. Environmental and genetics factors seem to have a complex interplay in genetically susceptible individuals leading to T1DM development.

Epigenetics is a new field of biology studying the inherited changes in deoxyribonucleic acid (DNA) expression which cannot be attributed to DNA sequence alteration via DNA methylation, histone modification, and micro-RNAs acting as post-transcriptional regulators.

The methylation of cytosine - guanosine dinucleotides (CpGs), located at the promoter region of the genes, play a vital role in transcription and gene expression and is catalyzed at the 5' cytosine position via enzymes called DNA methyltransferases (DNMTs).

A limited number of studies regarding epigenetics in T1DM paediatric patients have been published so far. The purpose of the present study is to investigate the CpG islet methylation pattern in the promoter regions of specific susceptibility genes such as Protein tyrosine phosphatase, non-receptor type 22 (PTPN-22), Insulin (INS) and Human leukocyte antigen G (HLA-G) genes, extracted from White Blood Cells (WBCs) from T1DM and healthy controls children and adolescents .

Twenty patients and twenty age and gender matched controls were recruited. A detailed personal, family, gestational/perinatal history was obtained and a thorough physical examination was performed in all study participants. Both groups and their first grade relatives had no history of other autoimmune diseases.

Parents provided written informed consent for the participation of their children, according to the declaration of Helsinki for research. involving human subjects .

Protocols were approved by Bioethics Committee of School of Medicine, Faculty of Health Sciences, Aristotle University of Thessaloniki, Thessaloniki, Greece (Protocol No 185/30.12.2015).

Whole blood samples were collected from both groups after a 12-hour period of fast and stored immediately at -80 oC.

DNA was extracted from blood samples using the DNA extraction kit QIAamp® DNA Blood Mini Kit (QIAGEN Inc, CA, USA), as suggested by the manufacturer. Isolated samples were quantified spectrophotometrically using the odds ratio (OD ratio) 260/280 (1 OD = 50 μg/ml), (BioPhotometer 6131 Eppendorf AG, Germany). Bisulfite-treatment was conducted on 300ng DNA of each sample by using the EZ DNA Methylation-Gold kit (Zymo Research, Methylation-Gold, USA), as recommended by the manufacturer. Treatment with sodium bisulphate converts unmethylated cytosines into uracils, whereas methylated cytosines remain unchanged under the same stable conditions.

For INS gene promoter amplification, gene-specific primers were used as follows: INS-Forward 5'-TATTTTGGAATTTTGAGTTTATT-3'and INS-Reverse 5'-AACAAAAATCTAAAAACAACAA-3', for PTPN-22-Forward 5'-TTTTGGTTTATGTTGTAGAGT -3΄ and PTPN-22 Reverse 5΄- ATTTTATTTTATTATTTATATGTAA-3' and for HLA-G- Forward 5'-TAGGGAGTTTAGTTTAGGGAT -3' and Reverse 5'- TTAAGGATGGTGGTTATGG -3'.

Additional, overhang adapter sequence was added to the locus-specific primers for the regions to be targeted (Nextera Transposase Adaptors, Illumina), in order of prompt construction of Next Generation Sequencing (NGS) libraries. Polymerase Chain Reaction (PCR) products were amplified on a low temperature ramping instrument, the 9700 thermal cycler (Eppendorf AG No5341, 9600 emulation mode) using the AmpliTaq Gold DNA Polymerase.

After purification of PCR products with highly reactive super magnetic beads NucleoMag NGS Clean-up and Size Select (Macherey-Nagel. Cat. Number 744970.5.), they were pooled at similar molar quantities and submitted for library construction according to manufacturer instructions, Nextera XT DNA Library Preparation kit, Research Illumina.

For NGS paired-end reads were selected at 2 x 250 base pair read length formation, on a platform Illumina's MiSeq.

Sequence analysis reads were carried out using FASTQ files and methylation status was estimated with the tool ampliMethProfiler, a python-based pipeline for targeted deep bisulfite sequenced amplicons.The methylation status was analyzed at ten CpG sites of INS gene promoter, four CpG sites of PTPN-22 gene and nineteen CpG sites of HLA-G gene around the transcriptional start site (TSS).

The sequences and the identification of the methylated and unmethylated sites will be interpreted by bioinformatics scientists.

A Data-Base will be created and all the data will undergo statistical analysis.The results and the conclusions of the present study will be published in peer- review journals and presented in National and International Meetings.

ELIGIBILITY:
Inclusion Criteria for both groups are:

* no history of T1DM or other autoimmune disease of their first degree relatives
* Greek origin (at least for 3 generations back to be Greek)
* sign written consent form

Inclusion Criteria for patients are:

* males and females 2-18 years of age, with the diagnosis of T1DM
* T1DM diagnosis according to the criteria of International Society for Pediatric and Adolescent Diabetes (ISPAD) and ADA (American Diabetes Association)

Inclusion Criteria for Controls are:

* healthy males and females 2-18 years of age, with no consaguinity with the patients

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents of Greek origin, aged 2-18 years old with a diagnosis of Type 1 Diabetes Mellitus as well as healthy controls age and gender matched.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Overall mean methylation percentage (%) of CpGs cytosine-guanosine islands within the promoter regions of INS, PTPN-22,HLA-G genes between T1DM and healthy children and adolescents | 5 years
  Calculation of the overall mean methylation percentage (%) of 10 cytosine-guanosine islands (CpGs) around the Transcription Start Site (TSS) of the INS gene promoter region, of 4 CpGs of PTPN-22 gene and of 19 CpG sites of HLA-G gene respectively between T1DM and control group

CONTACTS AND LOCATIONS:
Overall Officials: Assimina Galli-Tsinopoulou, MD,PhD, Principal Investigator — Unit of Pediatric Endocrinology/Diabetes/Metabolism 4thDepartment of Pediatrics
Locations (1):
- Unit of Pediatric Endocrinology, Diabetes and Metabolism-4th Department of Pediatrics, Medical School of Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu L, Li Y, Tollefsbol TO. Gene-environment interactions and epigenetic basis of human diseases. Curr Issues Mol Biol. 2008;10(1-2):25-36. PMID 18525104
- [Background] Dang MN, Buzzetti R, Pozzilli P. Epigenetics in autoimmune diseases with focus on type 1 diabetes. Diabetes Metab Res Rev. 2013 Jan;29(1):8-18. doi: 10.1002/dmrr.2375. PMID 23180441
- [Background] Barrett JC, Clayton DG, Concannon P, Akolkar B, Cooper JD, Erlich HA, Julier C, Morahan G, Nerup J, Nierras C, Plagnol V, Pociot F, Schuilenburg H, Smyth DJ, Stevens H, Todd JA, Walker NM, Rich SS; Type 1 Diabetes Genetics Consortium. Genome-wide association study and meta-analysis find that over 40 loci affect risk of type 1 diabetes. Nat Genet. 2009 Jun;41(6):703-7. doi: 10.1038/ng.381. Epub 2009 May 10. PMID 19430480
- [Background] Cooper JD, Simmonds MJ, Walker NM, Burren O, Brand OJ, Guo H, Wallace C, Stevens H, Coleman G; Wellcome Trust Case Control Consortium; Franklyn JA, Todd JA, Gough SC. Seven newly identified loci for autoimmune thyroid disease. Hum Mol Genet. 2012 Dec 1;21(23):5202-8. doi: 10.1093/hmg/dds357. Epub 2012 Aug 24. PMID 22922229
- [Background] Lu Q. The critical importance of epigenetics in autoimmunity. J Autoimmun. 2013 Mar;41:1-5. doi: 10.1016/j.jaut.2013.01.010. Epub 2013 Feb 1. PMID 23375849
- [Background] Quintero-Ronderos P, Montoya-Ortiz G. Epigenetics and autoimmune diseases. Autoimmune Dis. 2012;2012:593720. doi: 10.1155/2012/593720. Epub 2012 Mar 22. PMID 22536485
- [Background] Rakyan VK, Beyan H, Down TA, Hawa MI, Maslau S, Aden D, Daunay A, Busato F, Mein CA, Manfras B, Dias KR, Bell CG, Tost J, Boehm BO, Beck S, Leslie RD. Identification of type 1 diabetes-associated DNA methylation variable positions that precede disease diagnosis. PLoS Genet. 2011 Sep;7(9):e1002300. doi: 10.1371/journal.pgen.1002300. Epub 2011 Sep 29. PMID 21980303
- [Background] Saxonov S, Berg P, Brutlag DL. A genome-wide analysis of CpG dinucleotides in the human genome distinguishes two distinct classes of promoters. Proc Natl Acad Sci U S A. 2006 Jan 31;103(5):1412-7. doi: 10.1073/pnas.0510310103. Epub 2006 Jan 23. PMID 16432200
- [Background] Fradin D, Le Fur S, Mille C, Naoui N, Groves C, Zelenika D, McCarthy MI, Lathrop M, Bougneres P. Association of the CpG methylation pattern of the proximal insulin gene promoter with type 1 diabetes. PLoS One. 2012;7(5):e36278. doi: 10.1371/journal.pone.0036278. Epub 2012 May 2. PMID 22567146
- [Background] Grada A, Weinbrecht K. Next-generation sequencing: methodology and application. J Invest Dermatol. 2013 Aug;133(8):e11. doi: 10.1038/jid.2013.248. No abstract available. PMID 23856935
- [Background] Behjati S, Tarpey PS. What is next generation sequencing? Arch Dis Child Educ Pract Ed. 2013 Dec;98(6):236-8. doi: 10.1136/archdischild-2013-304340. Epub 2013 Aug 28. PMID 23986538
- [Background] Fisher MM, Watkins RA, Blum J, Evans-Molina C, Chalasani N, DiMeglio LA, Mather KJ, Tersey SA, Mirmira RG. Elevations in Circulating Methylated and Unmethylated Preproinsulin DNA in New-Onset Type 1 Diabetes. Diabetes. 2015 Nov;64(11):3867-72. doi: 10.2337/db15-0430. Epub 2015 Jul 27. PMID 26216854
- [Background] Lehmann-Werman R, Neiman D, Zemmour H, Moss J, Magenheim J, Vaknin-Dembinsky A, Rubertsson S, Nellgard B, Blennow K, Zetterberg H, Spalding K, Haller MJ, Wasserfall CH, Schatz DA, Greenbaum CJ, Dorrell C, Grompe M, Zick A, Hubert A, Maoz M, Fendrich V, Bartsch DK, Golan T, Ben Sasson SA, Zamir G, Razin A, Cedar H, Shapiro AM, Glaser B, Shemer R, Dor Y. Identification of tissue-specific cell death using methylation patterns of circulating DNA. Proc Natl Acad Sci U S A. 2016 Mar 29;113(13):E1826-34. doi: 10.1073/pnas.1519286113. Epub 2016 Mar 14. PMID 26976580
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Fisher MM, Perez Chumbiauca CN, Mather KJ, Mirmira RG, Tersey SA. Detection of islet beta-cell death in vivo by multiplex PCR analysis of differentially methylated DNA. Endocrinology. 2013 Sep;154(9):3476-81. doi: 10.1210/en.2013-1223. Epub 2013 Jul 3. PMID 23825129